CLINICAL TRIAL: NCT05933629
Title: Community-based Implementation of an Emotion Regulation Intervention for Individuals With Traumatic Brain Injury
Brief Title: Community-based Implementation of Online EmReg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Maria Kajankova, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-01380; 90DPTB0028-01-00 (Other Grant/Funding Number: National Institute On Disability & Rehabilitation Research)
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury; Emotion Regulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Training (Active Comparator): Participants assigned to this arm will complete a 3-hour training workshop on the intervention. After completing the training, participants will be asked to implement the intervention into their routine clinical practice.
  Interventions: Behavioral: Online EmReg
- Extended Training (Experimental): Participants assigned to this arm will complete the same 3-hour training workshop on the intervention as Arm #1. After completing the training, participants will also be asked to implement the intervention into their routine clinical practice. However, participants in this group will be asked to attend bi-weekly consultation sessions with members of the study team for 3 months following training.
  Interventions: Behavioral: Online EmReg; Behavioral: Consultation Sessions

INTERVENTIONS:
Behavioral: Online EmReg — A Web-based group intervention to improve emotion regulation in individuals with traumatic brain injury (TBI). Online EmReg is a 3-hour on-demand training workshop
Behavioral: Consultation Sessions — 3 months of bi-weekly consultation sessions
  Arms: Extended Training

SUMMARY:
This is a hybrid type III implementation-effectiveness trial; this study design blends elements of implementation and clinical effectiveness research, with the primary aim of determining the utility of an implementation strategy and a secondary aim of assessing clinical outcomes associated with the implementation trial. Consistent with best practices for this type of design, the study team will conduct a randomized test of the effect of implementation strategy on effective delivery of the Online EmReg intervention in clinical practice. Specifically, the study team will compare Standard Training (a 3-hour on-demand training workshop) to Extended Training, (a 3-hour on-demand training workshop with 3 months of bi-weekly consultation). The research team's primary aim is to determine the optimal strategy to train clinicians in effectively delivering Online EmReg, and secondary aim is to assess patient improvement per clinician-administered DERS. Outcome measures will be assessed via self-report surveys, performance evaluations (via role-plays), and tracked clinician participation and fidelity. Study participation is expected to last up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Licensed psychologist, social worker, or mental health counselor.
* Training and experience in CBT, the framework for EmReg.
* Experience working with people with TBI.
* Experience providing group treatment.
* A computer and internet to conduct group treatment via telehealth.
* Actively treating ≥3 patients with TBI who are appropriate for EmReg (have emotion regulation difficulties based on clinician assessment).
* Amenable to study tasks (e.g., completion of training, consultation, performance based role-play, data collection).
* Not previously trained in EmReg.
* Proficient in English.

Exclusion Criteria:

* Not willing to conduct group treatment via telehealth.
* Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Provider Self-Efficacy Scale Score | Up to 18 months
  A 7-item Likert Scale (not at all confident (1) to fully confident (7)) adapted for use with EmReg to assess provider confidence in delivering core components of the Online EmReg intervention. Total scores range from 26 to 182. Higher values indicate a higher level of self-efficacy. Used in the literature to reliably predict implementation of evidence-based interventions.
Performance Evaluation (via Role Plays) | Post-3 hour EmReg training workshop
  Assessed using a structured role play of EmReg groups in a simulated clinical setting. These role plays will be recorded and rated by a blinded evaluator. The evaluator will indicate the degrees to which the session goals were accomplished using a 15-item checklist. Each item will be rated a 0 (not introduced or covered), 1 (attempted/partially achieved), 2 (fully covered/achieved), or N/A (not applicable/relevant to session #). Participants can receive a total score of 0 to 30 on their performance-based role play. Higher values indicate higher achievement.

SECONDARY OUTCOMES:
Training Satisfaction Rating Scale | Up to 18 months
  Satisfaction with training will be assessed using the Training Satisfaction Rating Scale, a 12-item, 5-point Likert scale (higher scores = higher satisfaction). Total scores range from 12 to 60. Training engagement and consultation engagement (extended group only) will be tracked by study team.
Acceptability of Intervention Measure (AIM) | Up to 18 months
  Provider's satisfaction with the intervention will be assessed using the Acceptability of Intervention Measure (AIM), a 4-item, 5-point Likert scale. Total scores can range from 4 to 20 with higher scores indicating greater acceptability.
Feasibility of Intervention Measure (FIM) Scale | Up to 18 months
  Feasibility of the intervention will be assessed using the Feasibility of Intervention Measure (FIM), a 4-item, 5-point Likert scale. Total scores can range from 4 to 20 with higher scores indicating greater feasibility.
Intervention Appropriateness Measure (IAM) Scale | Up to 18 months
  Appropriateness of the intervention will be assessed using the Intervention Appropriateness Measure (IAM), a 4-item, 5-point Likert scale. Total scores can range from 4 to 20 with higher scores indicating greater intervention appropriateness.
Number of EmReg groups scheduled and completed | Up to 18 months
  The number of EmReg groups scheduled and completed by the clinician participants
Time between initial uptake and completion | Up to 18 months
  The time between completion of training and initial uptake will be tracked.
Skills Acquisition Quiz for Providers (SAQ-P) | Up to 18 months
  Clinician participants will be given a 25-item multiple-choice test of knowledge of Online EmReg training content. Correct answers are coded as 1 and incorrect answers are coded as 0. Scores range from 0-25 with higher scores indicating greater knowledge of the intervention.
Number of participants who receive treatment | Up to 18 months
  Clinician participants will be asked to track the number of patients who receive treatment out of those who appear eligible.
Difficulties in Emotion Regulation Scale (DERS) | Up to 18 months
  A 36-item questionnaire assessing capacity for emotion regulation. Each item is scored on a 5-point scale. Total scores range from 80 to 136. Out of the 36 items, 11 are reverse scored. Higher scores suggest greater problems with emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kajankova, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share individual participant data. Results will be published by the investigators in academic journals.